CLINICAL TRIAL: NCT06249984
Title: Effects of Tobacco Cut and Nicotine Form on the Abuse Liability of Moist Snuff
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brittney Keller-Hamilton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-22228; NCI-2023-01289 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K01DA055696 (NIH)
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Specimen Handling; Carbon Monoxide; Tobacco, Smokeless

STUDY DESIGN:
Intervention Model Description: Within-subjects factorial design
Who Masked: Participant
Masking Description: Blinded study products
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Prevention (Smokeless tobacco use: Usual Brand) (Placebo Comparator): Participants use their usual brand of moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Behavioral: Smokeless Tobacco Use; Other: Survey Administration
- Prevention (Smokeless tobacco use: Low FBN Long Cut) (Active Comparator): Participants use low FBN long cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Behavioral: Smokeless Tobacco Use; Other: Survey Administration
- Prevention (Smokeless tobacco use: Low FBN Fine Cut) (Active Comparator): Participants use low FBN fine cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Behavioral: Smokeless Tobacco Use; Other: Survey Administration
- Prevention (Smokeless tobacco use: High FBN Long Cut) (Active Comparator): Participants use high FBN long cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Behavioral: Smokeless Tobacco Use; Other: Survey Administration
- Prevention (Smokeless tobacco use: High FBN Fine Cut) (Active Comparator): Participants use high FBN fine cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Behavioral: Smokeless Tobacco Use; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Carbon Monoxide Measurement — Undergo CO test
  Other Names: Carbon Monoxide; CMONOX
Behavioral: Smokeless Tobacco Use — Use moist snuff
  Other Names: Tobacco, Smokeless
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests the effects of tobacco cut and nicotine form on the abuse liability in participants who use moist snuff (smokeless tobacco [SLT]). Two features of moist snuff that are key targets of manipulation from the tobacco industry and drivers of its addiction potential are length of tobacco cut (long versus fine) and nicotine form (low versus high levels of nicotine in the free-base form). Finer tobacco cuts and higher levels of free-base nicotine (FBN) result in faster, greater nicotine delivery. Researchers want to gain information on how certain characteristics of moist snuff affect how long people use it, how it delivers nicotine, or how much people like it. This clinical trial may provide justifications for local, state, or federal regulations aimed at reducing the appeal and addictiveness of moist snuff.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the association between style of moist snuff and SLT addiction among Ohio Appalachian adolescents and adults.

II. Characterize the carcinogen and free-base nicotine content of SLT products used by adolescents and adults with varying levels of SLT dependence in Ohio Appalachia.

III. Assess effects of moist snuff tobacco cut and FBN content on product use, effects, and appeal among Appalachian adults with high versus (vs.) low SLT dependence.

OUTLINE: Participants attend 5 study visits in a randomized order.

VISIT I: Participants use their usual brand of moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.

VISIT II: Participants use low FBN long cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.

VISIT III: Participants use low FBN fine cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.

VISIT IV: Participants use high FBN long cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.

VISIT V: Participants use high FBN fine cut moist snuff on study. Participants also undergo blood sample collection and carbon monoxide testing on study.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 (Adults Tobacco User Adult Cohort [TUAC]): Exclusive adult smokers who smoked >100 cigarettes or other combustible tobacco products in their lifetime and reported being current, every day, or some days/week smokers at time of enrollment
* AIM 1 (TUAC): Exclusive SLT user reporting every day or some days use per week at time of enrollment
* AIM 1 (TUAC): Or dual users who met criteria for both aims at time of enrollment who resided in participating Appalachian and urban counties
* AIM 1 (Buckeye Teen Health Study [BTHS]): Male youth ages 12-15 in Appalachian and urban regions of Ohio with parental consent and participant assent given
* AIM 2: As derived from Aim 1, commercially available SLT products used by TUAC and BTHS participants will be purchased from retailers in nearby Appalachian counties, as composition of SLT products can vary regionally
* AIM 3: Adults aged 21 and older who reside in Appalachian counties and surrounding rural areas under the RUCA code 10 classification and use SLT daily for at least 3 months and using 1.5 cans/week will be considered for this project
* Established moist snuff user (has used moist snuff daily for at least the past 3 months, uses at least 1.5 cans/week.
* Age 21 years or older
* Reside in Appalachian counties and surrounding rural areas under the RUCA code 10 classification
* Willing to complete 5 study visits and provide informed consent study procedures, including abstaining from all tobacco, nicotine, and marijuana for 12 hours before clinic visits
* Willing to abstain from nicotine and tobacco products 12-hours before study visit
* Ability to read and speak English

Exclusion Criteria:

* Pregnant, planning to become pregnant, or breastfeeding (will be verified with a urine pregnancy test at the first session visit)
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress, including but not limited to uncontrolled high blood pressure, chest pain, and shortness of breath, within the past 3 months
* Working with a cessation counselor, using cessation devices such as Chantix or Wellbutrin, or planning to quit within the next 3 months
* Severe periodontal or oral lesions

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequencies of flavors used by participants | Up to 2 years
  Will be assessed in adolescent and adult participants (expected N=198). Will be evaluated using descriptive statistics
Associations between tobacco cut (fine, long, and pouches) and level of smokeless tobacco (SLT) dependence | Up to 2 years
  Will use chi-square tests to estimate associations between tobacco cut (fine, long, and pouches) and level of SLT dependence. If the expected cell size for more than 20% of cells is < 5, Fisher's exact test will be used.
Associations between level of dependence and total nicotine in moist snuff | Up to 2 years
  Descriptive statistics will be calculated and variables will be inspected for out-of-range values. The investigators will merge product characteristics into our cohort study data (e.g., characteristics of Grizzly long cut wintergreen moist snuff will be merged to participants who reported using that style). Next, the investigators will use linear regression to estimate the associations between level of dependence and total nicotine.
Associations between level of dependence and pH in moist snuff | Up to 2 years
  Descriptive statistics will be calculated and variables will be inspected for out-of-range values. The investigators will merge product characteristics into our cohort study data (e.g., characteristics of Grizzly long cut wintergreen moist snuff will be merged to participants who reported using that style). Next, the investigators will use linear regression to estimate the associations between level of dependence and pH.
Associations between level of dependence and free-base nicotine (FBN) in moist snuff | Up to 2 years
  Descriptive statistics will be calculated and variables will be inspected for out-of-range values. The investigators will merge product characteristics into our cohort study data (e.g., characteristics of Grizzly long cut wintergreen moist snuff will be merged to participants who reported using that style). Next, the investigators will use linear regression to estimate the associations between level of dependence and FBN in moist snuff.
Moist snuff tobacco cut on product use | Up to 2 years
  Will be assessed by a randomized 2x2 within-subjects design to test whether variations in cut and level of FBN are associated with product use among Appalachian moist snuff users. Data will be summarized descriptively, overall and stratified by dependence. The investigators will use linear mixed effects models to assess the main effects of cut on moist snuff use duration and amount, self-reported measures, and plasma nicotine delivery (i.e., maximum absorption; total absorption; and speed of absorption). Product interaction terms will be used to evaluate whether effects of moist snuff style on outcome variables are modified by level of SLT dependence.
Moist snuff tobacco FBN content on product use | Up to 2 years
  Will be assessed by a randomized 2x2 within-subjects design to test whether variations in cut and level of FBN are associated with product use among Appalachian moist snuff users. Data will be summarized descriptively, overall and stratified by dependence. The investigators will use linear mixed effects models to assess the main effects of FBN content on moist snuff use duration and amount, self-reported measures, and plasma nicotine delivery (i.e., maximum absorption; total absorption; and speed of absorption). Product interaction terms will be used to evaluate whether effects of moist snuff style on outcome variables are modified by level of SLT dependence.
Moist snuff tobacco cut on product effects | Up to 2 years
  Will be assessed by a randomized 2x2 within-subjects design to test whether variations in cut and level of FBN are associated with subjective effects among Appalachian moist snuff users. Data will be summarized descriptively, overall and stratified by dependence. The investigators will use linear mixed effects models to assess the main effects of cut on moist snuff use duration and amount, self-reported measures, and plasma nicotine delivery (i.e., maximum absorption; total absorption; and speed of absorption). Product interaction terms will be used to evaluate whether effects of moist snuff style on outcome variables are modified by level of SLT dependence.
Moist snuff tobacco FBN content on product effects | Up to 2 years
  Will be assessed by a randomized 2x2 within-subjects design to test whether variations in cut and level of FBN are associated with subjective effects among Appalachian moist snuff users. Data will be summarized descriptively, overall and stratified by dependence. The investigators will use linear mixed effects models to assess the main effects of FBN content on moist snuff use duration and amount, self-reported measures, and plasma nicotine delivery (i.e., maximum absorption; total absorption; and speed of absorption). Product interaction terms will be used to evaluate whether effects of moist snuff style on outcome variables are modified by level of SLT dependence.
Moist snuff tobacco cut on product appeal | Up to 2 years
  Will be assessed by a randomized 2x2 within-subjects design to test whether variations in cut and level of FBN are associated with product use, nicotine delivery, and subjective effects among Appalachian moist snuff users. Data will be summarized descriptively, overall and stratified by dependence. The investigators will use linear mixed effects models to assess the main effects of cut on moist snuff use duration and amount, self-reported measures, and plasma nicotine delivery (i.e., maximum absorption; total absorption; and speed of absorption). Product interaction terms will be used to evaluate whether effects of moist snuff style on outcome variables are modified by level of SLT dependence.
Moist snuff tobacco FBN content on product appeal | Up to 2 years
  Will be assessed by a randomized 2x2 within-subjects design to test whether variations in cut and level of FBN are associated with product use, nicotine delivery, and subjective effects among Appalachian moist snuff users. Data will be summarized descriptively, overall and stratified by dependence. The investigators will use linear mixed effects models to assess the main effects of FBN content on moist snuff use duration and amount, self-reported measures, and plasma nicotine delivery (i.e., maximum absorption; total absorption; and speed of absorption). Product interaction terms will be used to evaluate whether effects of moist snuff style on outcome variables are modified by level of SLT dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Brittney L Keller-Hamilton, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Center for Tobacco Research, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu